CLINICAL TRIAL: NCT02856568
Title: A Phase Ib, Open-Label, Dose- Escalation Trial of ACY-1215 in Combination With Gemcitabine and Cisplatin in Patients With Unresectable or Metastatic Cholangiocarcinoma
Brief Title: Ricolinostat, Gemcitabine Hydrochloride, and Cisplatin in Treating Patients With Unresectable or Metastatic Cholangiocarcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Site dropped study
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1542; NCI-2016-01057 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1542 (Other: Mayo Clinic in Florida); P30CA015083 (NIH)
Record Dates: First submitted 2016-07-14; First posted 2016-08-05 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Non-Resectable Cholangiocarcinoma; Recurrent Cholangiocarcinoma; Stage III Extrahepatic Bile Duct Cancer; Stage III Intrahepatic Cholangiocarcinoma; Stage IIIA Hilar Cholangiocarcinoma; Stage IIIB Hilar Cholangiocarcinoma; Stage IVA Extrahepatic Bile Duct Cancer; Stage IVA Hilar Cholangiocarcinoma; Stage IVA Intrahepatic Cholangiocarcinoma; Stage IVB Extrahepatic Bile Duct Cancer; Stage IVB Hilar Cholangiocarcinoma; Stage IVB Intrahepatic Cholangiocarcinoma; Unresectable Extrahepatic Bile Duct Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms; Klatskin Tumor | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; ricolinostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cisplatin, gemcitabine hydrochloride, ricolinostat) (Experimental): Patients receive cisplatin IV followed by gemcitabine hydrochloride IV on days 1 and 8, and ricolinostat PO on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Ricolinostat

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloramine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Ricolinostat — Given PO
  Other Names: ACY-1215; Histone Deacetylase 6 InhibitorACY-1215

SUMMARY:
This phase Ib trial studies the side effects and best dose of ricolinostat when given together with gemcitabine hydrochloride and cisplatin in treating patients with cholangiocarcinoma that cannot be removed by surgery or has spread to other places in the body. Ricolinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine hydrochloride and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ricolinostat together with gemcitabine hydrochloride and cisplatin may work better in treating patients with cholangiocarcinoma that cannot be removed by surgery or has spread to other places.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) or a dose up to 240 mg/day, whichever is lower, of ricolinostat (ACY-1215) in combination with gemcitabine and cisplatin in patients with unresectable or metastatic cholangiocarcinoma. (Cohort I)

SECONDARY OBJECTIVES:

I. Characterize the safety profile of ACY-1215 in combination with gemcitabine and cisplatin in patients with unresectable or metastatic cholangiocarcinoma. (Both cohorts) II. Determine the single- and multiple-dose pharmacokinetic (PK) of ACY-1215 in combination with gemcitabine and cisplatin in patients with unresectable or metastatic cholangiocarcinoma. (Both cohorts) III. To evaluate tumor response to treatment with ACY-1215 in combination with gemcitabine and cisplatin (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria). (Both cohorts) IV. To assess progression-free and overall survival of patients treated with ACY-1215 in combination with gemcitabine and cisplatin. (Both cohorts)

TERTIARY OBJECTIVES:

I. Both blood and tissue samples will be obtained at baseline and post-treatment cycle 2 for future biomarker development, analysis, and potential blood based molecular/genomic profiling. (Both cohorts) II. Studies on Tissue pre-cycle 1 and post-cycle 2 of therapy will include: phospho extracellular signal-regulated kinases (ERK)1/2; hedgehog-signaling pathways (Gli transcription factors); BIM; histones acetylation; acetylation alpha (a)-tubulin; histone deacetylase (HDAC)6 levels; autophagy markers heat shock protein (HSP)90/70; hypoxia-inducible factor 1 (HIF1)alpha; beclin; microtubule-associated proteins 1A/1B light chain 3 (LC3); Ras homolog gene family member B (RhoB).

OUTLINE: This is a dose-escalation study of ricolinostat.

Patients receive cisplatin intravenously (IV) followed by gemcitabine hydrochloride IV on days 1 and 8, and ricolinostat orally (PO) on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytologic confirmation of unresectable or metastatic cholangiocarcinoma (intrahepatic, hilar, extrahepatic bile duct)
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Absolute neutrophil count (ANC) >= 1200/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin < 1.5 x upper limit of normal (ULN), If patient has known Gilbert's syndrome, direct bilirubin < 2.0 x ULN
* Aspartate transaminase (AST) =< 5 x ULN
* Alkaline phosphatase =< 5 x ULN
* Creatinine =< 1.5 x ULN
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Ability to complete a patient medication diary by themselves or with assistance
* Provide informed written consent
* Willingness to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willingness to provide tissue and blood samples for correlative research purposes
* Life expectancy >= 3 months
* Prior embolization, chemoembolization, or radiofrequency ablation permitted if >= 4 weeks from registration and evidence of new tumor growth is present

Exclusion Criteria:

* Any of the following

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Central nervous system (CNS) metastasis; NOTE: history of brain metastasis other than locally treatable lesions (i.e., lesions treatable with surgery or radiosurgery); patients with locally treatable disease may be considered for study if they have completed treatment without evidence of CNS progression for > 4 weeks after completion of treatment; patients with a history of brain or other CNS metastases not amenable to local therapy will not be eligible
* Prior biologic or immunologic therapy =< 4 weeks prior to study entry
* Prior systemic chemotherapy for cholangiocarcinoma or gallbladder carcinoma; NOTE: adjuvant chemotherapy is allowed if completed > 6 months prior to the start of registration
* Prior radiation of cholangiocarcinoma or gallbladder carcinoma; NOTE: adjuvant radiation therapy is allowed if completed > 6 months prior to the start of registration
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 5 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix or breast, or prostatic intraepithelial neoplasm; NOTE: if there is a history or prior malignancy, patient must not be receiving other specific treatment (other than hormonal therapy) for their cancer
* History of myocardial infarction =< 6 months from registration, or congestive heart failure requiring use of ongoing maintenance therapy for life threatening ventricular arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
MTD of ricolinostat or a dose up to 240 mg/day whichever is lower, of ACY-1215 | Cycle 1, Day 1 pre-dose
  PK blood sample
MTD of ricolinostat or a dose up to 240 mg/day whichever is lower, of ACY-1215 | Cycle 1, Day 8 pre-dose
  PK blood sample
MTD of ricolinostat or a dose up to 240 mg/day whichever is lower, of ACY-1215 | 0.5 hr after ACY-1215 dosing
  PK blood sample
MTD of ricolinostat or a dose up to 240 mg/day whichever is lower, of ACY-1215 | 24 hr after Cycle 1, Day 1 only
  PK blood sample
MTD of ricolinostat or a dose up to 240 mg/day whichever is lower, of ACY-1215 | Prior to Cycle 1, Day 2 ACY-1215 dosing
  PK blood sample
MTD of ricolinostat or a dose up to 240 mg/day whichever is lower, of ACY-1215 | 1 hr after ACY-1215 dosing
  PK blood sample
MTD of ricolinostat or a dose up to 240 mg/day whichever is lower, of ACY-1215 | 2hr after ACY-1215 dosing
  PK blood sample
MTD of ricolinostat or a dose up to 240 mg/day whichever is lower, of ACY-1215 | 4 hr after ACY-1215 dosing
  PK blood sample
MTD of ricolinostat or a dose up to 240 mg/day whichever is lower, of ACY-1215 | 6-8 hr after ACY-1215 dosing
  PK blood sample

SECONDARY OUTCOMES:
Best Response defined as the best objective status recorded using RECIST version 1.1 | Up to 1 year
  Responses will be summarized by simple descriptive summary statistics.
Confirmed response is defined to be a stringent complete response, complete response, very good partial response, or partial response noted as the objective status on two consecutive evaluations using RECIST version 1.1 | Up to 1 year
  Will be evaluated using all cycles of treatment. Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group). The number of responses may indicate further evaluation for specific tumor types in a Phase II setting.
Incidence of adverse events evaluated via the ordinal common toxicity criteria (CTC) toxicity grading of 3+ | Up to 1 year
  Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Time to any hematologic nadirs (ANC, platelets, hemoglobin) | Up to 1 year
  Will be summarized descriptively.
Time to any treatment related grade 3+ toxicity | Up to 1 year
  Will be summarized descriptively.
Time to any treatment related toxicity | Up to 1 year
  Will be summarized descriptively.
Time to progression | From registration to documentation of progression, up to 1 year
  Will be summarized descriptively.
Time to treatment failure | From registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient assessed up to 1 year
  Will be summarized descriptively.

OTHER OUTCOMES:
Laboratory correlates measured from tissue by western blot | Up to 1 year
  Descriptive statistics and simple scatterplots will form the basis of presentation of these data. Correlations between these laboratory values and other outcome measures like response will be carried out in an exploratory manner.
Laboratory correlates measured from tissue by immunofluorescence | Up to 1 year
  Descriptive statistics and simple scatterplots will form the basis of presentation of these data. Correlations between these laboratory values and other outcome measures like response will be carried out in an exploratory manner.

CONTACTS AND LOCATIONS:
Overall Officials: Kabir Mody, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota